CLINICAL TRIAL: NCT04248634
Title: Short and Midterm Results of Delayed Colo-anal Anastomosis After Rectal Resection
Brief Title: Evaluation of Delayed Coloanal Anastomosis
Acronym: ACAD
Status: Completed | Type: Observational
Sponsor: Institut National d'Oncologie, Morocco (Other Government)
Responsible Party: Principal Investigator, Anass Majbar, Professor of surgery, Institut National d'Oncologie, Morocco
Other Study IDs: SCOD 1
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Rectal Neoplasms
Keywords: Rectal neoplasmdelayed coloanal anastomosis; Ileostomy; Delayed coloanal anastomosis
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Delayed colo-anal anastomosis — Colo-anal anastomosis performed in two surgical steps:
  - Step one: the colon is exteriorized transanally and 5 cm of the colon is left outside without anastomosis creation.
  Step two: after 7 days, the excess colon is resected and the colo-anal anastomosis is created.

SUMMARY:
After rectal resection for cancer of the lower rectum, the restoration of continuity is done by a colo-anal anastomosis with a protective ileostomy. However, the ileostomy is very little accepted by patients. It is associated with significant morbidity and a deterioration in the quality of life.

Delayed colo-anal anastomosis has been proposed as an alternative to direct colo-anal anastomosis with a protective ileostomy. The theoretical advantage of this technique is to reduce the risk of anastomotic leaks and to avoid ileostomy.

In this study, the investigators will retrospectively evaluate the short and midterm results of this technique.

DETAILED DESCRIPTION:
After rectal resection for cancer of the lower rectum, the restoration of continuity is done by a colo-anal anastomosis with a protective ileostomy. The latter reduces the risk and severity of clinical anastomotic fistulas. However, the ileostomy is very little accepted by patients. It is associated with significant morbidity reaching up to 30% of patients, a deterioration in the quality of life and the need for a second surgery to restore digestive continuity. And specifically in low-income countries, ostomy bags are expensive and are not reimbursed, and therefore constitute a heavy burden for Moroccan patients.

In order to overcome these drawbacks, delayed colo-anal anastomosis has been proposed as an alternative to direct colo-anal anastomosis with a protective ileostomy. This technique consists of externalizing the colon in the first stage by the transanal route, without creating an ileostomy, and waiting a week for the creation of the anastomosis. The theoretical advantage of this technique is to reduce the risk of anastomotic leaks and to avoid ileostomy. Several studies have shown encouraging results in the short and midterm, and it is listed among the technical options in the French recommendations for the management of rectal cancer.

In this study, the investigators will retrospectively evaluate the short and midterm results of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients> 18 years old.
* Rectal resection with the creation of a delayed colo-anal anastomosis.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients aged above 18 years, who undergo rectal resection with the creation of delayed colo-anal anastomosis.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Stoma rate at 90 days | 90 days
  The rate of patients who required a stoma creation at 90 days
Perineal complications | 90 days
  Rates of perineal complications at 90 days after surgery

SECONDARY OUTCOMES:
Clavien-Dindo complications | 90 days
  Rate of complications according to Clavien-Dindo grading
Functional outcomes | 12 months
  Continence score according to the Low anterior resection syndrom score (LARS). Score from 0 to 42 (0-20 No LARS / 21-29 Minor LARS / 30-42 Major LARS). Higher score indicates worse outcome
Quality of life assessement: EORTC QLQ30 score | 12 months
  Quality of life using the EORTC QLQ30 score at 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut National d'Oncologie, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: Undecided
Under reasonable request, we would share individual patient dara